CLINICAL TRIAL: NCT06442046
Title: Strengthening the Connections to Opportunities for Prevention Engagement (SCOPE)
Brief Title: Strengthening the Connections to Opportunities for Prevention Engagement
Acronym: SCOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kevin Borrup (Other)
Collaborators: The Tow Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Kevin Borrup, Executive Director, Injury Prevention Center, Connecticut Children's Medical Center
Organization: Connecticut Children's Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-052
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Interpersonal Violence; Structural Violence
Keywords: youth violence prevention
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Enrolled subjects will provide the study team with email, mobile, work phone, physical contact address, and contact numbers for two or more close contacts. Families will be contacted monthly by the case manager assist with additional supports they might need. Quarterly, patients and families will be contacted and patients will be asked to complete VPET and other measures. The intervention group will receive active case management to connect affected youth to community services.
  Interventions: Other: Active Case Management; Other: Treatment as usual
- Treatment as Usual (Active Comparator): The comparison group will receive treatment as usual which consists of a list of community resources and a recommendation that youth not already connected with a community service provider be connected.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Active Case Management — A case manager will work with families post-discharge to ensure that youth are connected to an appropriate community support. Case managers will also work with families to identify any social needs and provide support in accessing services as needed.
  Arms: Intervention
Other: Treatment as usual — Subjects will receive a list of youth serving community service agencies and provided a recommendation to connect to them.

SUMMARY:
The Strengthening the Connections to Opportunities for Prevention Engagement (SCOPE) project will create a pathway for children and families from the City of Hartford to connect with a Connecticut Children's Care Coordinator (CC) in an effort to reduce levels of violence exposure.

DETAILED DESCRIPTION:
The Strengthening the Connections to Opportunities for Prevention Engagement (SCOPE) project will create a pathway for children and families from the City of Hartford to connect with a Connecticut Children's Care Coordinator (CC) when they are determined to have high levels of violence exposure.

SCOPE seeks to decrease future violence exposure and increase resiliency of children with high levels of exposure to violence through Emergency Department (ED)-based case management and connections with community partners.

Hypothesis 1: VPET scores within the intervention group will show significant reductions across the study period. The percent of patients with positive VPET positive scores within the intervention group will show significant reductions from the expected 79% to 70% as compared to the control group that will have the expected 79%

Hypothesis 2: The Child and Youth Resilience Measure-Revised (CYRM) scores for the intervention group will increase by 10%, and will be significantly higher than the control group.

Hypothesis 3: At least 75% of the intervention group will be assessed as "positive" for having made a connection with community services.

Hypothesis 4: 90% of parents with children receiving case management will report being satisfied with the case management services and community connected services.

Hypothesis 5: Retention within the intervention group will be at or above 50%, with at least half of participants remaining engaged in the project.

Hypothesis 6: Compared to the control group, the intervention group will have fewer documented injuries and ED visits during the 12-month period post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

* At least 8 years of age and not older than 17 years of age (until 18th birthday)
* Hartford resident based on zip code of primary residence or parent report?
* Accompanied by a parent or guardian who can provide consent
* Capable of providing assent/consent
* Able to provide consent in English or Spanish
* Presenting at CT Children's during recruitment hours

Exclusion Criteria:

* Patients whose primary complaint is for behavioral health
* Patients in Connecticut Department of Children and Families (DCF) or police custody

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 225 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline violence exposure at 12 months | Baseline and months 3, 6, 9, and 12
  A reduction in exposure as measured using the Violence Prevention Emergency Tool (VPET) that provides a range from 0 to 21 with a 4 or more considered elevated.

SECONDARY OUTCOMES:
Change in resilience score from baseline at 12 months | Baseline and months 3, 6, 9, and 12
  The Child and Youth Resilience Measure-Revised (CYRM) is a validated scale with resilience scores that range from 17 to 85 with a higher score indicating greater resilience.
Difference in connections between intervention and control at 3-month intervals. | Quarterly measure at 0, 3, 6, 9, and 12 months
  A dichotomous yes/no variable answering the question of are you currently connected to services at a community agency?
Level of satisfaction with case management services after 12 months of services | At 12-months of case management.
  Level of satisfaction with case management services as indicated along a 5-point scale from Not satisfied to Completely satisfied. Higher levels of satisfaction are related with other improved outcomes from baseline.
Rate of re-injury in the intervention group compared to the control condition. | baseline, 3, 6, 9, 12 months
  Hospital documented injuries during the study period will be assessed on a quarterly schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Borrup, DrPH, Principal Investigator — Connecticut Children's
Locations (1):
- Connecticut Children's, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No